CLINICAL TRIAL: NCT04601532
Title: Randomized Controlled Trial Assessing a Novel Glycopolymer Compound in the Treatment of Superficial Partial-thickness Burns
Brief Title: Superficial Partial-Thickness Burn Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Delayed recruitment
Sponsor: J. Peter Rubin, MD (Other)
Collaborators: Synedgen, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, J. Peter Rubin, MD, Endowed Chair of Plastic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20050205
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Superficial Partial Thickness Burn
MeSH Terms: interventions — Silver Sulfadiazine

STUDY DESIGN:
Intervention Model Description: This study is an investigator initiated, single site, University of Pittsburgh, prospective, parallel group, randomized controlled trial comparing SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel (intervention group) to the current gold standard treatment Silvadene (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Silver sulfadiazine (Active Comparator): Topical management via dressings provide a barrier against microbial infection. The current gold standard for burn wound dressings is silver (nanoparticulate or ionic), and it has shown some efficacy in treating infections, but it does not demonstrate an ability to prevent infections and some treatment guidelines even recommend against its use. Although silver dressing is preferred for military use, a retrospective review spanning 10 years of use in military environments showed that silver was not more effective than other antimicrobial topical treatments, and a meta-analysis with over 2500 surgical patients found silver sulfadiazine was associated with increased infection rates and hospital length-of-stays were two days longer on average.
  Interventions: Drug: Silver Sulfadiazine
- Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser (Experimental): Synedgen has developed Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser. These products are Food and Drug Administration (FDA) 510(k) cleared wound care medical devices, formulated with a novel biocompatible chitosan derivative, poly (acetyl, arginyl) glucosamine. SynePure™ Wound Cleanser is optimized for the cleansing and debridement of wounds and thermal injuries, and Catasyn™ Advanced Technology Hydrogel serves as a protective gel dressing. Together, these products reduce inflammation in wounds, aggregate bacteria and disrupt bacterial biofilms, and accelerate healing.
  Interventions: Device: Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser

INTERVENTIONS:
Device: Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser — Catasyn™ Advanced Technology Hydrogel is a wound hydrogel that provides a moist wound environment. A moist wound environment is supportive to wound healing. SynePure™ Wound Cleanser is a non-cytotoxic wound cleanser for the removal of foreign material from epidermal and dermal wounds, burns, cuts, abrasions and minor irritations of the skin.
  Arms: Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Drug: Silver Sulfadiazine — Silver sulfadiazine, a sulfa drug, is used to prevent and treat infections in burn wounds.
  Other Names: Silvadene Topical Product
  Arms: Silver sulfadiazine

SUMMARY:
This study is an investigator initiated, single site, University of Pittsburgh, prospective, parallel group, randomized controlled trial comparing SynePure Wound Cleanser and Catasyn Advanced Technology Hydrogel (intervention group) to the current gold standard treatment Silvadene (control group). Both groups will receive the same care other than the treating agent. Subjects will be recruited form the UPMC Mercy Burn Center adult patient pool who have sustained superficial partial-thickness burn wounds that comprise less than or equal to 10% of total body surface area (TBSA)

DETAILED DESCRIPTION:
Current effective dressings for burn wounds contain silver (nanoparticulate or ionic), hypochlorite, hydrogen peroxide, sulfa agents, chlorhexidine, iodine or other dilute antiseptics meant to provide some measure of antimicrobial protection. However, all of these materials have some proven limitations in facilitating wound healing and also have notable local and systemic adverse effects. None of the current clinical treatments enhance healing and/or reduce scar formation. The purpose of this study is to test the safety and effectiveness of SynePure™ Wound Cleanser when used in combination with Catasyn™ Advanced Technology Hydrogel for the treatment of superficial partial-thickness burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* 18 years of age or older, male and female
* Patients who have sustained superficial, partial-thickness burn wounds ≤ to 10% of total body surface area (TBSA)
* Patients otherwise in good general physical and mental health, as per the investigator's clinical judgment

Exclusion Criteria:

* Inability to provide informed consent
* Deep partial-thickness burns and full-thickness burns
* Radiation, chemical, or electrical burn injury
* Patients with burns primarily located to the face, genitals, or span across joints
* Patients whose burn injury was ≥ to 48 hours prior to entry into the UPMC Mercy Burn Center Clinic.
* Patients with uncontrolled cerebrovascular disease, cardiovascular disease, endocrine disease, hepatic disease, or renal disease; or other severe conditions for whom, in the physician investigators' discretion, would render study participation unsafe
* Patients with documented or self-reported shellfish allergies
* Current pregnancy
* Patients with concurrent burn related injuries or inhalation injury that would put the patient at increased risk, per physician discretion
* Any condition to which in the investigator's discretion would render study enrollment a safety concern for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Mercy Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Church D, Elsayed S, Reid O, Winston B, Lindsay R. Burn wound infections. Clin Microbiol Rev. 2006 Apr;19(2):403-34. doi: 10.1128/CMR.19.2.403-434.2006. PMID 16614255
- [Background] Duran N, Duran M, de Jesus MB, Seabra AB, Favaro WJ, Nakazato G. Silver nanoparticles: A new view on mechanistic aspects on antimicrobial activity. Nanomedicine. 2016 Apr;12(3):789-799. doi: 10.1016/j.nano.2015.11.016. Epub 2015 Dec 24. PMID 26724539
- [Background] Aziz Z, Abu SF, Chong NJ. A systematic review of silver-containing dressings and topical silver agents (used with dressings) for burn wounds. Burns. 2012 May;38(3):307-18. doi: 10.1016/j.burns.2011.09.020. Epub 2011 Oct 24. PMID 22030441
- [Background] Aurora A, Beasy A, Rizzo JA, Chung KK. The Use of a Silver-Nylon Dressing During Evacuation of Military Burn Casualties. J Burn Care Res. 2018 Jun 13;39(4):593-597. doi: 10.1093/jbcr/irx026. PMID 29901799
- [Background] Barajas-Nava LA, Lopez-Alcalde J, Roque i Figuls M, Sola I, Bonfill Cosp X. Antibiotic prophylaxis for preventing burn wound infection. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD008738. doi: 10.1002/14651858.CD008738.pub2. PMID 23740764
- [Background] Wasiak J, Cleland H. Burns: dressings. BMJ Clin Evid. 2015 Jul 14;2015:1903. PMID 26173045
- [Background] Narayanaswamy VP, Giatpaiboon SA, Uhrig J, Orwin P, Wiesmann W, Baker SM, Townsend SM. In Vitro activity of novel glycopolymer against clinical isolates of multidrug-resistant Staphylococcus aureus. PLoS One. 2018 Jan 17;13(1):e0191522. doi: 10.1371/journal.pone.0191522. eCollection 2018. PMID 29342216
- [Background] Narayanaswamy VP, Keagy LL, Duris K, Wiesmann W, Loughran AJ, Townsend SM, Baker S. Novel Glycopolymer Eradicates Antibiotic- and CCCP-Induced Persister Cells in Pseudomonas aeruginosa. Front Microbiol. 2018 Aug 3;9:1724. doi: 10.3389/fmicb.2018.01724. eCollection 2018. PMID 30123191
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734
- [Background] Oliveira GV, Chinkes D, Mitchell C, Oliveras G, Hawkins HK, Herndon DN. Objective assessment of burn scar vascularity, erythema, pliability, thickness, and planimetry. Dermatol Surg. 2005 Jan;31(1):48-58. doi: 10.1111/j.1524-4725.2005.31004. PMID 15720096
- [Background] Li-Tsang CW, Lau JC, Liu SK. Validation of an objective scar pigmentation measurement by using a spectrocolorimeter. Burns. 2003 Dec;29(8):779-84. doi: 10.1016/s0305-4179(03)00165-7. PMID 14636751
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Background] Maruish M. User's manual for the SF-12v2 Health Survey. 3. Lincoln, RI: QualityMetric Inc.; 2012.
- [Background] Cheak-Zamora NC, Wyrwich KW, McBride TD. Reliability and validity of the SF-12v2 in the medical expenditure panel survey. Qual Life Res. 2009 Aug;18(6):727-35. doi: 10.1007/s11136-009-9483-1. Epub 2009 May 8. PMID 19424821
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Elliott D; Bluebelle Study Group. Developing outcome measures assessing wound management and patient experience: a mixed methods study. BMJ Open. 2017 Nov 26;7(11):e016155. doi: 10.1136/bmjopen-2017-016155. PMID 29180591
- [Background] Nherera L, Trueman P, Roberts C, Berg L. Silver delivery approaches in the management of partial thickness burns: A systematic review and indirect treatment comparison. Wound Repair Regen. 2017 Aug;25(4):707-721. doi: 10.1111/wrr.12559. Epub 2017 Aug 17. PMID 28742235

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawn due to allergic reaction to Silver sulfadiazine. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Please see participant flow for details of subject withdraw and lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 9 | 9 | 18
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
The patient and observer scar assessment scale (POSAS) [Mean (Full Range); unit: Mean Total POSAS Baseline Score] — The patient and observer scar assessment scale (POSAS) is used to measure scar quality. It is composed of a patient reported section and an observer reported section (6 scored items each). Each section consists of items on a ten-step scale (1= as normal skin to 10=very different from normal skin/worst scar imaginable). A higher score indicates more symptoms/issues present; the lower the score the closer to normal skin. These are then summed together to make up the total score (maximum of 120 and minimum of 12).
  Mean Total POSAS Baseline Score | 64 [17 to 108] | 65 [26 to 107] | 64 [17 to 108]

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Healing of the Superficial Partial Thickness Burn Wound.
Description: Number of days to healed burn wound (re-epithelialization as defined by greater than or equal to 90% epithelialized wound, determined by investigator exam and review of wound photographs, as needed)
Time Frame: up to 21 days
Population: 23 subjects completed the study. Two subjects in the SynePure+ Catasyn group were lost-to-follow-up, and one subject in the silver sulfadiazine group withdrew due to an adverse reaction. Additionally, one subject missed three study visits (37.5% of visits) but did complete the first and final visits, so the primary outcomes were still available. All 26 subjects received at least one treatment and were included in the intention-to-treat analysis.
Measure: Median (Full Range); unit: Days to healing
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
Days to healing | 7 [7 to 11.5] | 9 [7.5 to 18]

2. Primary Outcome: Change From Screening Visit to Visit 8 in Total Patient and Observer Scar Assessment Scale (POSAS) Score
Description: The patient and observer scar assessment scale (POSAS) is used to measure scar quality. It is composed of a patient reported section and an observer reported section (6 scored items each). Each section consists of items on a ten-step scale (1= as normal skin to 10=very different from normal skin/worst scar imaginable). A higher score indicates more symptoms/issues present; the lower the score the closer to normal skin. These sections are then summed together to make up the total score (maximum of 120 and minimum of 12). Please note the means listed denote the difference in POSAS score between the baseline and last assessment completed (21 days if last visit completed, or earlier visit if withdrawn or lost to follow up).
Time Frame: up to 21 days
Population: The sample size was too small to perform the planned analysis with confidence that the results are valid and represent the population (total n = 26, n = 13 per group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
score on a scale | 29.9 (10.5) | 30.5 (12.5)

3. Secondary Outcome: Safety- Infection Rate From Screening Visit to Visit 8
Description: Safety as measured by total incidences of infection from screening visit to visit 8, or to last visit completed, for the three lost to follow up participants, and 1 participant who was withdrawn.
Time Frame: up to 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

4. Secondary Outcome: Safety- Rate of Noted Wound Progression From Screening Visit to Visit 8
Description: Safety as measured by total incidence of progression of burn wounds to deep partial thickness/full thickness from screening visit to visit 8, or to last visit completed, for the three lost to follow up participants, and 1 participant who was withdrawn.
Time Frame: up to 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

5. Secondary Outcome: Safety- Rate of Complications From Screening Visit to Visit 8
Description: Safety as measured by rate of adverse event/complication that resulted in a change to the participant's treatment course from initial standard of care from screening visit to visit 8, or to last visit completed, for the three lost to follow up participants, and 1 participant who was withdrawn.
Time Frame: up to 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
Participants | 1 | 0

6. Secondary Outcome: Safety- as Measured by Change in Total Vancouver Scar Scale Score From Screening Visit to Visit 8, or to Last Visit Completed, for the Three Lost to Follow up Participants, and 1 Participant Who Was Withdrawn.
Description: Vancouver Scar Scale Score: The VSS is a scale to assess the extent of scarring for a given wound by scoring the pigmentation, vascularity, pliability and height of the scar. Each domain is individually scored then the domains are summed to give a total score that range from zero (0) to 13 with zero (0) representing a 'normal' presentation. Validity and reliability of the scale have been documented and is commonly used in wound healing research. The means listed represent the difference in total score from baseline to 21 days, or from baseline to last assessment, if participant did not complete the 21 day visit.
Time Frame: up to 21 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
Number analyzed (Participants) | 13 | 13
score on a scale | 3.6 (2.3) | 3.2 (1.6)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Silver Sulfadiazine | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver Sulfadiazine (N=13) | Catasyn™ Advanced Technology Hydrogel and SynePure™ Wound Cleanser (N=13)
Burn to left shoulder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild, unrelated to study procedure or product.
Bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Mild, unrelated to study procedure or product.
Dermal budding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild, unrelated to study procedure or product.
Limb swelling (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Mild, unrelated to study procedure or product.
pain (burning/stinging) (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (4) — Mild, unrelated to study procedure or product.
Parathesis, tingling (Nervous system disorders) | 1 (1) | 1 (1) — Mild, unrelated to study procedure or product.
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild, unrelated to study procedure or product.
Warmth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild, unrelated to study procedure or product.
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild, unrelated to study procedure or product.
headache (General disorders) | 1 (1) | 0 (0) — Mild, unrelated to study procedure or product.
Sinusitis (General disorders) | 1 (1) | 0 (0) — Mild, unrelated to study procedure or product.
Skin rash, allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild, probably related to study product (silver sulfadiazine). Per PI, subject was withdrawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04601532/Prot_SAP_ICF_000.pdf